CLINICAL TRIAL: NCT06658431
Title: Study on Music Intervention of Non-clinical College Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ye Zhiyin (Other)
Responsible Party: Sponsor-Investigator, Ye Zhiyin, Teaching assistant, Central University of Finance and Economics, China
Organization: Central University of Finance and Economics, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUFE2
Record Dates: First submitted 2024-10-20; First posted 2024-10-26 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-10

CONDITIONS: Depression Anxiety Disorder
Keywords: music therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): 90 minutes music group therapy
  Interventions: Behavioral: music group therapy
- control group (No Intervention): Without any intervention

INTERVENTIONS:
Behavioral: music group therapy — 90 minutes music group therapy
  Arms: Experimental group

SUMMARY:
The purpose of this trial is to understand whether a mindfulness-integrated volleyball team sports program can effectively intervene in the mental health of college students. The main questions it aims to answer is:

Does the music group effectively intervene in the participants' mental health levels, including indicators such as anxiety and depression?

Participants will:

Attend a music group once a week for 1.5 hours each session, for a total of 6 weeks.

Complete a psychological questionnaire every 3 weeks and a follow-up questionnaire every 2 weeks after the program concludes for twice.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 16 years or older.
* Able to communicate in Mandarin and voluntarily participate in the study.
* Agree to consistently participate in each session.

Exclusion Criteria:

* Disagree to consistently participate in each mindfulness-integrated volleyball course.
* Individuals unable to commit to participating in each mindfulness-integrated volleyball course.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
depression | From enrollment to 4 weeks after the end of treatment.
  Using GAD-7 to investigate the psychological variables of participants, a total of four assessments will be conducted, including T1 pre-test (before the start), with measurement time points at T2 (after 3 weeks of intervention), T3 (after 6 weeks of intervention), T4 (2 weeks after the end)， and T5 (4 weeks after the end).
anxiety | From enrollment to 4 weeks after the end of treatment.
  Using PHQ-9 to investigate the psychological variables of participants, a total of four assessments will be conducted, including T1 pre-test (before the start), with measurement time points at T2 (after 3 weeks of intervention), T3 (after 6 weeks of intervention), T4 (2 weeks after the end) and T5 (4 weeks after the end).
perceived stress | From enrollment to 4 weeks after the end of treatment.
  Using PSS-10 to investigate the psychological variables of participants, a total of four assessments will be conducted, including T1 pre-test (before the start), with measurement time points at T2 (after 3 weeks of intervention), T3 (after 6 weeks of intervention), T4 (2 weeks after the end) and T5 (4 weeks after the end).

SECONDARY OUTCOMES:
sleep | From enrollment to 4 weeks after the end of treatment.
  Using ISI-7 to investigate the psychological variables of participants, a total of four assessments will be conducted, including T1 pre-test (before the start), with measurement time points at T2 (after 3 weeks of intervention), T3 (after 6 weeks of intervention), T4 (2 weeks after the end) and T5 (4 weeks after the end).
positive and negative affective | From enrollment to 4 weeks after the end of treatment.
  Using PANAS-10 to investigate the psychological variables of participants, a total of four assessments will be conducted, including T1 pre-test (before the start), with measurement time points at T2 (after 3 weeks of intervention), T3 (after 6 weeks of intervention), T4 (2 weeks after the end) and T5 (4 weeks after the end).
life satisfaction | From enrollment to 4 weeks after the end of treatment.
  Using SWLS-5 to investigate the psychological variables of participants, a total of four assessments will be conducted, including T1 pre-test (before the start), with measurement time points at T2 (after 3 weeks of intervention), T3 (after 6 weeks of intervention), T4 (2 weeks after the end) and T5 (4 weeks after the end).
burnout | From enrollment to 4 weeks after the end of treatment.
  Using MBI-SS-15 to investigate the psychological variables of participants, a total of four assessments will be conducted, including T1 pre-test (before the start), with measurement time points at T2 (after 3 weeks of intervention), T3 (after 6 weeks of intervention), T4 (2 weeks after the end) and T5 (4 weeks after the end).
emotion regulation | From enrollment to 4 weeks after the end of treatment.
  Using ERQ-10 to investigate the psychological variables of participants, a total of four assessments will be conducted, including T1 pre-test (before the start), with measurement time points at T2 (after 3 weeks of intervention), T3 (after 6 weeks of intervention), T4 (2 weeks after the end) and T5 (4 weeks after the end).
loneliness and social anxiety | From enrollment to 4 weeks after the end of treatment.
  Using UCLA Scale to investigate the psychological variables of participants, a total of four assessments will be conducted, including T1 pre-test (before the start), with measurement time points at T2 (after 3 weeks of intervention), T3 (after 6 weeks of intervention), T4 (2 weeks after the end) and T5 (4 weeks after the end).
self acceptance | From enrollment to 4 weeks after the end of treatment.
  Using SAQ-16 to investigate the psychological variables of participants, a total of four assessments will be conducted, including T1 pre-test (before the start), with measurement time points at T2 (after 3 weeks of intervention), T3 (after 6 weeks of intervention), T4 (2 weeks after the end) and T5 (4 weeks after the end).
perceived support | From enrollment to 4 weeks after the end of treatment.
  Using MSPSS-6 to investigate the psychological variables of participants, a total of four assessments will be conducted, including T1 pre-test (before the start), with measurement time points at T2 (after 3 weeks of intervention), T3 (after 6 weeks of intervention), T4 (2 weeks after the end) and T5 (4 weeks after the end).

CONTACTS AND LOCATIONS:
Locations (1):
- Central University of Finance and Economics, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided